CLINICAL TRIAL: NCT02093312
Title: Meals on Wheels, a Randomized Controlled Study on the Effect of a Home Food-delivery Service for Cancer Patients
Brief Title: Meals on Wheels, the Effect of a Home Food-delivery Service for Cancer Patients
Acronym: RUMLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Christian Bitz, Head of Reseach, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EFFECT.A03.2014
Record Dates: First submitted 2014-02-20; First posted 2014-03-21 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Lung Cancer; Ambulant; Malnourished
Keywords: Cancer; Food-delivery; Nutritional Intervention; Quality of life; Outpatients
MeSH Terms: conditions — Lung Neoplasms; Malnutrition; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): The control group is not offered any home food-delivery service, but continues with their habitual diet
- Intervention group (Experimental): The intervention group is offered home food-delivery service
  Interventions: Dietary Supplement: Home food-delivery service

INTERVENTIONS:
Dietary Supplement: Home food-delivery service — A home food-delivery service is offered the intervention group of cancer patients
  Arms: Intervention group

SUMMARY:
The overall objective of the study is to investigate the effect of energy- and protein enriched home delivered meals vs. habitual diet in malnourished patients suffering from cancer on various endpoints.

DETAILED DESCRIPTION:
Despite the fact that nutritional deterioration has been associated with patients' functional impairment, the effect of individualized nutritional support or counselling to outpatients, focussing on ordinary food, have not yet been thoroughly explored (Ravasco P. et al. 2007). A few studies have investigated the effect of nutritional counselling on quality of life (QoL) in cancer patients after discharge (Ovesen et al. 1993, Persson et al. 2002, Isenring et al. 2004, Ravasco et al. 2005a, Ravasco et al. 2005b). However, there is to our knowledge not conducted any studies examining the effect of home delivered meals on QoL and other endpoints in outpatients suffering from cancer.

The overall objective of the study is to measure the effect of energy- and protein enriched home delivered meals vs. habitual diet in malnourished outpatients diagnosed with lung cancer. The intervention diet will consist of optional protein- and energy-dense main and in-between-meals. There will be 22 different main meals and 13 in-between meals to choose between. The meals are prepared by The Nordic Kitchen of Copenhagen University Hospital Herlev. The offered main meals will consist of a selection of warm dishes taken from the ordinary menu. The in-between meals are a collection of the Delights of Herlev (dishes previously shown to increase dietary intake among in-patients). The food will be delivered to the participants' home 3 times per week, and participants can order one warm dish and ad libitum in-between meals for each day.

ELIGIBILITY:
Inclusion Criteria:

* Have a nutritional risk score ≥ 3 according to NRS-2002 (Kondrup J. et al. 2003)
* Be diagnosed with lung cancer
* Have a life expectancy > 12 weeks
* Not plan to loose weight or go on a diet
* Not plan to go on vacation for > 2 weeks during the study period
* Live at their own home
* Live ≤ 25 km from the hospital
* Be able to read, write and understand Danish

Exclusion Criteria:

* Receives food from a food-delivery service
* Have food allergies or intolerance
* Exclusively receives enteral or parenteral nutrition
* Suffers from cognitive impairment e.g. dementia
* Is terminal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6 weeks (change from baseline)
  To assess the Global QoL, a questionnaire from the European Organization for the Research and Treatment of Cancer (EORTC) QLQ-30, version 3, will be used. This is a validated, cancer-specific questionnaire with a total of 30 questions, looking back at the past week. The scoring of QoL is based on 2 specific questions with response options ranging from 1-7 which indicate very bad to very good. A Danish version of the questionnaire will be used.
Quality of Life | 12 weeks (change from baseline)
  To assess the Global QoL, a questionnaire from the European Organization for the Research and Treatment of Cancer (EORTC) QLQ-30, version 3, will be used. This is a validated, cancer-specific questionnaire with a total of 30 questions, looking back at the past week. The scoring of QoL is based on 2 specific questions with response options ranging from 1-7 which indicate very bad to very good. A Danish version of the questionnaire will be used.

SECONDARY OUTCOMES:
Hand grip strength | 6, and 12 weeks (changes from baseline)
  Hand grip strength (in kg) will be measured with a Hydraulic Hand Dynamometer. Participants will be seated with forearms rested on the arms of the chair. They are asked to perform three maximum force trials with their dominant hand and using the second handle position. The test will be repeated within 30 seconds, and the maximum grip score from the three measured values will be used.
30-second chair-stand test | 6, and 12 weeks (changes from baseline)
  The 30-second-chair-stand test consist of manually counting the number of sit-stand-sit cycles completed during the 30 seconds of the test. A standard chair (with a seat height of 40cm) with or without a backrest but with armrests will be used. Initially, subject will be seated on the chair with their back in an upright position. They will be instructed to rise after the "1, 2, 3, go" command at their own preferred speed with their arms folded across their chest. If the participant is only able to perform the test by using armrest, the test will be recorded as "modified".
Body Weight | 6, and 12 weeks (changes from baseline)
  Body weight will be measured to the nearest 0.1 kg following standard procedures (i.e. without shoes, minimal clothing).
Depression Scale | 6, and 12 weeks (changes from baseline)
  The Center for Epidemiological Studies Depression scale (CES-D) is a short self-report scale designed to measure depressive symptoms (Hann D. et al. 1999). The questionnaire contains 20 items, divided in four domains: Somatic Retarded Activity (7 items), Depressed Affect (5 items), Positive Affect (4 items), and Interpersonal Affect (2 items), and 2 single items that complete the total score. The total score ranges from 0 to 60; a score of ≥16 indicates a depressed symptomatology. The CES-D has been validated in several samples of cancer patients, and it is often administered to inpatients with cancer (Vodermaier A. et al. 2009). A Danish version of the questionnaire will be used.
Total energy- and protein intake per day | 6, and 12 weeks (changes from baseline)
  Dietary intake will be assessed by a dietary interview covering patient's dietary intake over the past week. On basis of the dietary interview the total energy and protein intake per day is estimated. A food database with energy- and protein content of various foods is used for the estimation.
Re-admissions with total length of stay (LOS) | 12 weeks, and 6 months
  Data on re-admissions to the hospital and LOS will be collected from all participants medical charts (hospital medical system OPUS/GS).
Mortality | 12 weeks, and 6 months
  Data on mortality will be collected from all participants' medical charts (hospital medical system OPUS/GS).
WHO Performance status | 6, and 12 weeks
Functional-score | 6 and 12 weeks
  Using EORTC-QLQ-30 version 3 - looking back at the past week. Out of the 30 questions the functional score is based on 15 specific questions with 4 response options indicating either: not at all, a little, some or a lot. Involves questions related to physical-, role-, emotional-, cognitive- and social functioning.
Symptom-score | 6 and 12 weeks (changes from baseline)
  Using EORTC-QLQ-30 version 3 - looking back at the past week. Out of the 30 questions the symptom score is based on 13 specific questions with 4 response options indicating either: not at all, a little, some or a lot.

OTHER OUTCOMES:
Compliance | 1, 6, and 12 weeks
  All patients in the intervention group are requested to daily fulfil a compliance sheet during the whole 12-week period, where the intake of intervention dishes will be recorded. Project staff will review the completed sheets together with the study participant at mid-way (week 6) and at the final 12-week visit in order to minimize possible uncertainties. Moreover, eventual side-effects and reasons for non-compliance will be recorded.
Evaluation | 12 weeks
  All the intervention participants will receive an evaluation form in order to assess the acceptability of the offered meals, the food-delivery service, and a possible price they would give for this particular food-delivery service.
Effect of social status on total energy- and protein intake | Baseline
  Definition of social status: if the participant is living alone or not
Correlation between compliance (intervention group) and Quality of life | 12 weeks
Correlation between total energy- and protein intake (all participants) and Quality of life | 12 weeks
Correlation between compliance (intervention group) and Body weight | 12 weeks
Correlation between compliance (intervention group) and Hand grib strength | 12 weeks
Correlation between compliance (intervention group) and 30-second chair-stand test | 12 weeks
Correlation between compliance (intervention group) and Depression score | 12 weeks
Correlation between compliance (intervention group) and Total energy- and protein intake | 12 weeks
Correlation between compliance (intervention group) and WHO performance status | 12 weeks
Correlation between total energy- and protein intake (all participants) and Hand grip strength | 12 weeks
Correlation between total energy- and protein intake (all participants) and Body weight | 12 weeks
Correlation between total energy- and protein intake (all participants) and 30 second chair-stand test | 12 weeks
Correlation between total energy- and protein intake (all participants) and Depression scale | 12 weeks
Correlation between total energy- and protein intake (all participants) and WHO performance status | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arne V Astrup, Professor, Principal Investigator — University of Copenhagen; Eva Leedo, Cand Scient, Study Director — University of Copenhagen
Locations (1):
- Herlev University Hsopital, Herlev, Denmark

REFERENCES:
- [Result] Leedo E, Gade J, Granov S, Mellemgaard A, Klausen TW, Rask K, Astrup A. The Effect of a Home Delivery Meal Service of Energy- and Protein-Rich Meals on Quality of Life in Malnourished Outpatients Suffering from Lung Cancer: A Randomized Controlled Trial. Nutr Cancer. 2017 Apr;69(3):444-453. doi: 10.1080/01635581.2017.1283421. Epub 2017 Feb 17. PMID 28287324